CLINICAL TRIAL: NCT01901640
Title: Phase 3 Study to Evaluate Longterm Safety of Once-a-Day Dosing of Udenafil in the Treatment of Erectile Dysfunction
Brief Title: Safety Study of Once-a-Day Dosing of Udenafil to Treat Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA8159_EDDL_III
Record Dates: First submitted 2013-01-22; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DA-8159 (Experimental): Udenafil(The study had one arm.)
  Interventions: Drug: DA-8159 (Udenafil)

INTERVENTIONS:
Drug: DA-8159 (Udenafil)

SUMMARY:
Phase : Phase III Indication : Erectile Dysfunction Study Design : open-label, fixed dose, 6-month extension study (parent study : DA8159_EDD_III)

DETAILED DESCRIPTION:
Completer from parent study(DA8159_EDD_III)continued into a 24weeks open-label extension during which they received udenafil once daily. The study concluded with a 4-week ED treatment-free period.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 20 years or more diagnosed with erectile dysfunction(ED)

Exclusion Criteria:

* Had uncontrolled blood pressure
* Had hepatic or renal dysfunction
* Had significant psychiatric disorders or drug abuses
* Was currently under anticancer chemotherapy
* Had a treatments for ED using other phosphodiesterase type 5(PDE-5) inhibitors

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety | 48 weeks(after 24 weeks of parent study), 52weeks(after 28weeks of parent study)
  Safety evaluation included adverse events, standard 12-lead electrocardiograms and clinical laboratory measures. The AEs measured as percentage and number of patients.

SECONDARY OUTCOMES:
International Index of Erectile Function(IIEF), GAQ(Global Assessment Questions), Shift to normal | 48 weeks(after 24 weeks of parent study), 52weeks(after 28weeks of parent study)
  The efficacy measures(Unit of Measure)
  * IIEF EF domain score(Change from baseline)
  * IIEF other domain scores(Change from baseline)
  * GAQ & Shift to normal(percentage of subject)

CONTACTS AND LOCATIONS:
Overall Officials: S W Kim, MD, PhD, Principal Investigator — the Catholic University of Korea St. Mary's Hospital; D G Moon, MD, PhD, Principal Investigator — Korea University Guro Hospital; J J Kim, MD, PhD, Principal Investigator — Korea University Anam Hospital; N C Park, MD, PhD, Principal Investigator — Pusan National University Hospital; S W Lee, MD, PhD, Principal Investigator — Samsung Medical Center; J S Paick, MD, PhD, Principal Investigator — Seoul National University Hospital; T Y Ahn, MD, PhD, Principal Investigator — Asan Medical Center; K H Moon, MD, PhD, Principal Investigator — Yeungnam University Hospital; W S Chung, MD, PhD, Principal Investigator — Ewha Womans University Hospital; K S Min, MD, PhD, Principal Investigator — Inje University; J K Park, MD, PhD, Principal Investigator — Chonbuk National University Hospital; D Y Yang, MD, PhD, Principal Investigator — Kangdong Sacred Heart Hospital